CLINICAL TRIAL: NCT00290355
Title: A Phase IIB Study to Assess the Efficacy of GSK 249553 as Adjuvant Therapy Given to MAGE-3-Positive Patients With Non-Small-Cell Lung Cancer in Stage IB (T2/N0) or II (T1/N1 or T2/N1 or T3/N0), Who Have Had Complete Surgical Resection
Brief Title: Study to Test the Efficacy of the Vaccine GSK 249553 in Treating Non-small-cell Lung Cancer After Tumour Removal by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 249553/004
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2019-02-25 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer, Non-Small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GSK 249553 Group (Experimental): Male and female patients at least 18 years of age, with resectable non-small-cell lung cancer (NSCLC), who received 13 doses of GSK 249553 vaccine, administered intramuscularly in the deltoid or lateral regions of the thighs, alternatively on the right and left sides, according to the following schedule: 5 doses at 3-week intervals, followed by 8 doses at 3-month intervals.
  Interventions: Biological: GSK 249553 vaccine
- Placebo Group (Placebo Comparator): Male and female patients at least 18 years of age, with resectable non-small-cell lung cancer (NSCLC), who received 13 doses of placebo, administered intramuscularly in the deltoid or lateral regions of the thighs, alternatively on the right and left sides, according to the following schedule: 5 doses at 3-week intervals, followed by 8 doses at 3-month intervals.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GSK 249553 vaccine — Intramuscular injection, 13 doses
  Arms: GSK 249553 Group
Biological: Placebo — Intramuscular administration, 13 doses
  Arms: Placebo Group

SUMMARY:
Patients will receive injections of GSK 249553 vaccine . Appropriate tests will be performed to assess the safety of the treatment and its ability to induce an immune response.

DETAILED DESCRIPTION:
This Phase IIb study will be conducted at centres in several European countries according to a multicentre, international, randomised, double-blind design. It will provide information about the clinical and immunological efficacy and the tolerability of GSK 249553 when this is administered to patients with stage IB, II NSCLC. The study treatment will be administered by intramuscular injection; first administration will take place 4-6 weeks after surgery. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained prior to surgical tumour resection and prior to the performance of any other protocol-specific procedures.
* At least 18 years of age at the time of resection.
* Pathologically proven, surgically staged squamous or non-squamous IB, IIA or IIB NSCLC, and complete surgical resection.
* The operative technique for resection of the patient's tumour involves at least a lobectomy or a sleeve lobectomy, conforming to all of the following criteria:

  1. Removal of all gross disease with negative resection margins, by lobectomy, sleeve resection, bilobectomy or pneumonectomy, based on intra-operative findings.
  2. The level of nodal sampling is at least as follows:

Levels 4, 7, 10 in both right upper and right middle lobes Levels 4, 7, 9, 10 in right lower lobe Levels 5, 6, 7 in left upper lobe Levels 7, 9, 10 in left lower lobe. or at the maximum defined as systematic radical mediastinal lymphadenectomy: all ipsilateral and easily accessible lymph-node levels must be removed, independently of the location of the primary tumour. The level of nodal sampling is as follows: Levels 2, 4, 7, 8, 9, 10 in right-sided tumours, Levels 5, 6, 7, 8, 9, 10 in left-sided tumours

* Tumour shows expression of MAGE-3 antigen.
* Recovered from surgery for at least 4 weeks and not more than 6 weeks.
* ECOG performance status of ≤ 1 at the time of randomisation.
* Laboratory criteria (all of the following must be fulfilled): adequate bone marrow reserve, adequate renal function, adequate hepatic function, serum bilirubin within normal range, negative HIV antibody test, negative HBV antigen test, negative HCV antibody test.
* (For females): EITHER not of child-bearing potential OR sexually abstinent OR all of the following: negative urine/serum β-HCG pregnancy test, use of adequate contraceptive precautions for 30 days before first vaccination. Agree to continue such precautions for 2 months after completion of the course of vaccination.

Exclusion Criteria:

* Received any anti-cancer specific treatment including radiotherapy, prior to surgery, unless the treatment was for previous malignancies allowed by the protocol, i.e., basal and localised squamous-cell skin carcinoma that has been successfully treated, or carcinoma in situ of the cervix (see exclusion criterion no. 10).
* Candidate for post-surgery radiation therapy or any kind of anti-cancer-specific treatment.
* Pregnant/lactating.
* (For female patients of child-bearing potential): not agree to practice an effective method of contraception.
* Uncontrolled bleeding disorder.
* Autoimmune disease.
* History of anaphylaxis or severe allergic reaction.
* Undergone splenectomy or radiation to the spleen.
* Received a major organ allograft.
* Malignancies at other sites (except (i) basal and localised squamous-cell skin carcinoma that has been successfully treated, and (ii) carcinoma in situ of the cervix).
* Concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* Uncontrolled congestive heart failure or hypertension.
* Unstable heart disease or uncontrolled arrhythmia at the time of enrolment.
* Psychiatric or addictive disorders that may compromise ability to give informed consent, or to comply with the trial procedures.
* Any evidence of residual tumour after surgery.
* Require concomitant treatment with systemic corticosteroids, or any other immunosuppressive agents.
* Received chemotherapy, immunotherapy related to NSCLC.
* Need home oxygenation.
* Received any investigational or non-registered drug or vaccine other than the study vaccine within the 30 days preceding the first dose of study vaccine, or plans to receive such a drug during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2002-05-28 (Actual); Primary Completion 2011-07-19 (Actual); Study Completion 2011-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (59):
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (2):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Tampere
- France (2):
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Rennes
- Germany (18):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Villingen-Schwenningen, Baden-Wurttemberg
  - GSK Investigational Site, Ebensfeld, Bavaria
  - GSK Investigational Site, Gauting, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Offenbach, Hesse
  - GSK Investigational Site, Delmenhorst, Lower Saxony
  - GSK Investigational Site, Hemer, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Kaiserslautern, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Bad Berka, Thuringia
  - GSK Investigational Site, Berlin
- Greece (3):
  - GSK Investigational Site, Marousi
  - GSK Investigational Site, Rio-Patras
  - GSK Investigational Site, Thessaloniki
- Italy (5):
  - GSK Investigational Site, Pordenone, Friuli Venezia Giulia
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Perugia, Umbria
  - GSK Investigational Site, Venezia, Veneto
- Latvia (2):
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Rigas Rajons
- GSK Investigational Site, Vilnius, Lithuania
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Nijmegen
- Norway (2):
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Trondheim
- Poland (6):
  - GSK Investigational Site, Chęciny
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Tuszyn
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Zakopane
- Spain (7):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Valencia
- United Kingdom (2):
  - GSK Investigational Site, Hull
  - GSK Investigational Site, London
- GSK Investigational Site

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=4970

REFERENCES:
- [Background] Passlick B et al. MAGE-A3 Antigen-Specific Cancer Immunotherapeutic (ASCI) as adjuvant therapy in resected stage IB/II Non-Small Cell Lung Cancer (NSCLC): from proof-of-concept to Phase III trial (MAGRIT). Abstract presented at the European Multidisciplinary Conference in Thoracic Oncology (EMCTO), Lugano, Switzerland. 1-3 May 2009; 64 (suppl. 1):S45 (102PD).
- [Background] Vansteenkiste J et al. Activity of MAGE-A3 cancer immunotherapeutic as adjuvant therapy in stage IB/II Non-Small Cell Lung Cancer (NSCLC): Final results of a multi-center, double-blind, randomized, placebo-controlled Phase II study. Abstract presented at the 12th Conference on Lung Cancer (WCLC), Seoul, Korea. 2-6 September 2007.
- [Background] Vansteenkiste J et al. Adjuvant therapy in stage IB/II Non-Small Cell Lung Cancer (NSCLC): Final results of a multi-center, double-blind, randomized, placebo-controlled Phase II study evaluating the MAGE-A3 cancer immunotherapeutic. Abstract presented at The 14th European Cancer Conference (ECCO) (formerly ECCO14/ESTRO 26), Barcelona, Spain. 23-27 September 2007.
- [Background] Vansteenkiste J et al. Multi-center, double-blind, randomized, placebo-controlled Phase II study to assess the efficacy of recombinant MAGE-A3 vaccine as adjuvant therapy in stage IB/II MAGE-A3-positive, completely resected, Non-Small Cell Lung Cancer (NSCLC). Abstract presented at the 43rd Annual Meeting American Society of Clinical Oncology (ASCO), Chicago, IL. 1-5 June 2007.
- [Background] Vansteenkiste J et al. Multi-center, double-blind, randomized, placebo-controlled phase II study to assess the efficacy of recombinant MAGE-A3 vaccine as adjuvant therapy in stage IB/II MAGE-A3-positive, completely resected, non-small-cell lung cancer (NSCLC). Abstract presented at the 42nd Annual Meeting American Society of Clinical Oncology (ASCO), Atlanta, GA. 2-6 June 2006.
- [Background] Vansteenkiste J et al. Phase II randomized study of MAGE-A3 immunotherapeutic as adjuvant therapy in stage IB/II Non-Small Cell Lung Cancer (NSCLC): 44 month follow-up, humoral and cellular immune response data. European Society for Medical Oncology (IASLC-ESMO) Abstract presented at the 1st European Lung Cancer Conference (ELCC), Geneva, Switzerland. 23-26 April 2008; 3 (4 suppl.1):S55-56.
- [Background] Zielinski M et al. MAGE-A3 Antigen-Specific Cancer Immunotherapeutic (ASCI) as adjuvant therapy in resected stage IB/II Non-Small Cell Lung Cancer (NSCLC): from proof-of-concept to Phase III trial (MAGRIT). Abstract presented at the 17th European Conference on General Thoracic Surgery (ECGTS), Krakow, Poland. 31 May-3 June 2009.
- [Derived] Zhu J, Yuan Y, Wan X, Yin D, Li R, Chen W, Suo C, Song H. Immunotherapy (excluding checkpoint inhibitors) for stage I to III non-small cell lung cancer treated with surgery or radiotherapy with curative intent. Cochrane Database Syst Rev. 2021 Dec 6;12(12):CD011300. doi: 10.1002/14651858.CD011300.pub3. PMID 34870327
- [Derived] Vansteenkiste J, Zielinski M, Linder A, Dahabreh J, Gonzalez EE, Malinowski W, Lopez-Brea M, Vanakesa T, Jassem J, Kalofonos H, Perdeus J, Bonnet R, Basko J, Janilionis R, Passlick B, Treasure T, Gillet M, Lehmann FF, Brichard VG. Adjuvant MAGE-A3 immunotherapy in resected non-small-cell lung cancer: phase II randomized study results. J Clin Oncol. 2013 Jul 1;31(19):2396-403. doi: 10.1200/JCO.2012.43.7103. Epub 2013 May 28. PMID 23715567
- [Derived] Ulloa-Montoya F, Louahed J, Dizier B, Gruselle O, Spiessens B, Lehmann FF, Suciu S, Kruit WH, Eggermont AM, Vansteenkiste J, Brichard VG. Predictive gene signature in MAGE-A3 antigen-specific cancer immunotherapy. J Clin Oncol. 2013 Jul 1;31(19):2388-95. doi: 10.1200/JCO.2012.44.3762. Epub 2013 May 28. PMID 23715562
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 249553/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 249553/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 249553/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 249553/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 249553/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 249553/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 249553/004 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK 249553 Group | Placebo Group
Started | 122 | 60
Completed | 105 | 55
Not Completed | 17 | 5
Not completed — Serious adverse event | 7 | 4
Not completed — Study product reactogenicity | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Migrated / moved from the study area | 1 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK 249553 Group | Placebo Group | Total
Number analyzed (Participants) | 122 | 60 | 182
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (7.85) | 62.6 (8.88) | 62.53 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 23
  Male | 106 | 53 | 159
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 122 | 60 | 182

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reporting Confirmed Non-small-cell Lung Cancer (NSCLC) Recurrence
Description: Types of recurrence included local, regional and distant metastasis and second primary lung tumours, and comprised: Local recurrence, defined as a tumour within the same lung or at the bronchial stump; Regional recurrence, involving a clinically or radiologically manifest disease in the mediastinum or in supraclavicular nodes; and Distant recurrence, i.e., any tumour arising in the contralateral lung or outside the hemithorax. The time to recurrence was defined as the interval from the date of surgical resection to the date of recurrence. The latter was defined as the date of the first study assessment at which new lesion(s) were found and confirmed by appropriate imaging.
Time Frame: Over a median follow-up time of 28 months post-Dose 1
Population: The analyses were performed on the Total Treated cohort, which included all patients who were randomised and who received at least one dose of the randomised study product administration. This analysis was based on the confirmed NSCLC recurrence so that patients withdrawn before imaging were removed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 114 | 57
Participants | 37 | 24
Statistical Analysis 1: Comparison: GSK 249553 Group vs Placebo Group; Hazard ratio of GSK 249553 study product; Test type: Other; p = 0.256, Regression, Cox — Two-sided p value from Cox regression model adjusted for covariate(s) node/squam/stage to test the null hypothesis was: the distribution of time to recurrences was the same in each group (H0 = [HR=1]); The p value by log rank test was 0.1995. Criterion for evaluation of the objective: one sided p-value < 10%; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.44 to 1.24]

2. Secondary Outcome: Percentage of Patients With Disease Recurrence
Description: as for outcome 1
Time Frame: At 6, 12, 18, 24 and 30 months after enrolment
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 114 | 57
Percentage of Patients
  Recurrence at Month 6 | 89.1 | 91.5
  Recurrence at Month 12 | 78.6 | 70.8
  Recurrence at Month 18 | 72.4 | 62.0
  Recurrence at Month 24 | 68.8 | 58.3
  Recurrence at Month 30 | 63.8 | 58.3

3. Secondary Outcome: Number of Patients Reporting Confirmed Non-small-cell Lung Cancer (NSCLC) Recurrence or Death - Disease Free Survival (DFS)
Description: as for outcome 1
Time Frame: Over a median follow-up time of 44 months post-Dose 1
Population: The analyses were performed on the Total Treated cohort, which included all patients who were randomised and who received at least one dose of the randomised study product administration.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 122 | 60
Participants | 49 | 29

4. Secondary Outcome: Number of Participants Who Died - Overall Survival (OS)
Description: Overall Survival (OS) was based on total number of deaths, irrespective of cause of death. Non-small-cell Lung Cancer Overall Survival (NSCLC-OS) was based on total number of deaths due to lung cancer; deaths due to other or to unknown causes were censored appropriately.
Time Frame: Over a median follow-up time of 44 months post-Dose 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 122 | 60
Participants
  Deaths, any cause | 36 | 21
  Deaths, NSCLC-related | 27 | 13

5. Secondary Outcome: Number of Subjects Seropositive Against MAGE-A3
Description: A seropositive subject was defined as a subject whose antibody concentration was greater than or equal to (≥) 27.000 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Day 0, Week 6, Week 12, Month 9, Month 18, Month 24, at Month 30 and at Follow-Up (FU) visit (Post Dose 13 at Month 42 for patients with full treatment course or Post last product dose + 12 months for the other patients)
Population: The analyses were performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable patients for whom immunogenicity post product administration data were available for the considered assay. For each patient, data collected after major protocol violation were eliminated from ATP immunogenicity analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 119 | 57
Participants
  Day 0 | 9 | 6
  Week 6: number analyzed (Participants) | 110 | 54
  Week 6 | 88 | 4
  Week 12: number analyzed (Participants) | 100 | 47
  Week 12 | 98 | 5
  Month 9: number analyzed (Participants) | 76 | 34
  Month 9 | 75 | 2
  Month 18: number analyzed (Participants) | 56 | 26
  Month 18 | 56 | 2
  Month 24: number analyzed (Participants) | 52 | 23
  Month 24 | 52 | 1
  Month 30: number analyzed (Participants) | 44 | 20
  Month 30 | 44 | 2
  FU visit: number analyzed (Participants) | 27 | 6
  FU visit | 25 | 1

6. Secondary Outcome: Anti- MAGE-A3 Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 119 | 57
EL.U/mL
  Day 0 | 16.9 [14.4 to 19.8] | 17.8 [13.8 to 23.0]
  Week 6: number analyzed (Participants) | 110 | 54
  Week 6 | 120.1 [88.1 to 163.6] | 17.0 [13.4 to 21.5]
  Week 12: number analyzed (Participants) | 100 | 47
  Week 12 | 1017.4 [793.6 to 1304.4] | 18.7 [13.8 to 25.2]
  Month 9: number analyzed (Participants) | 76 | 34
  Month 9 | 505.9 [404.1 to 633.3] | 14.7 [13.0 to 16.6]
  Month 18: number analyzed (Participants) | 56 | 26
  Month 18 | 673.7 [508.0 to 893.6] | 14.7 [13.0 to 16.6]
  Month 24: number analyzed (Participants) | 52 | 23
  Month 24 | 627.5 [464.8 to 847.1] | 14.0 [13.0 to 15.0]
  Month 30: number analyzed (Participants) | 44 | 20
  Month 30 | 783.0 [571.8 to 1072.2] | 14.8 [12.9 to 16.8]
  FU visit: number analyzed (Participants) | 27 | 6
  FU visit | 187.8 [118.4 to 297.9] | 16.1 [10.2 to 25.4]

7. Secondary Outcome: Number of Subjects Seropositive Against Protein D (PD) Antigens
Description: A seropositive subject was defined as a subject whose antibody concentration was greater than or equal to (≥) 100.000 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 115 | 55
Participants
  Day 0 | 45 | 16
  Week 6: number analyzed (Participants) | 110 | 51
  Week 6 | 100 | 19
  Week 12: number analyzed (Participants) | 99 | 47
  Week 12 | 99 | 20
  Month 9: number analyzed (Participants) | 75 | 28
  Month 9 | 75 | 12
  Month 18: number analyzed (Participants) | 56 | 25
  Month 18 | 56 | 11
  Month 24: number analyzed (Participants) | 52 | 23
  Month 24 | 52 | 7
  Month 30: number analyzed (Participants) | 43 | 20
  Month 30 | 43 | 8
  FU visit: number analyzed (Participants) | 26 | 7
  FU visit | 26 | 0

8. Secondary Outcome: Anti-protein D (Anti-PD) Antibody Concentrations
Description: as for outcome 6
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 115 | 55
EL.U/mL
  Day 0 | 92.2 [78.6 to 108.0] | 71.6 [60.9 to 84.2]
  Week 6: number analyzed (Participants) | 110 | 51
  Week 6 | 711.7 [539.4 to 939.1] | 78.9 [65.6 to 94.8]
  Week 12: number analyzed (Participants) | 99 | 47
  Week 12 | 2694.0 [2179.6 to 3329.9] | 87.7 [71.6 to 107.5]
  Month 9: number analyzed (Participants) | 75 | 28
  Month 9 | 1455.8 [1137.0 to 1864.0] | 88.3 [65.9 to 118.4]
  Month 18: number analyzed (Participants) | 56 | 25
  Month 18 | 2029.0 [1591.2 to 2587.1] | 85.9 [64.0 to 115.3]
  Month 24: number analyzed (Participants) | 52 | 23
  Month 24 | 1587.7 [1197.2 to 2105.5] | 78.9 [55.4 to 112.4]
  Month 30: number analyzed (Participants) | 43 | 20
  Month 30 | 2018.4 [1486.6 to 2740.4] | 78.8 [59.3 to 104.6]
  FU visit: number analyzed (Participants) | 26 | 7
  FU visit | 812.6 [513.9 to 1284.9] | 50.0 [50.0 to 50.0]

9. Secondary Outcome: Number of Subjects With Cell-mediated Immunity (CMI) Cluster of Differentiation (CD) 4+ Response
Description: Responders were patients with at least 5x10-⁶ increase in minimal CD4 precursor frequency versus baseline. Any = at least one post treatment time point.
Time Frame: At Week 6, Week 12, Month 9, Month 18, Month 24, at Month 30 and at Follow-Up (FU) visit (Post Dose 13 at Month 42 for patients with full treatment course or Post last product dose + 12 months for the other patients)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 37 | 14
Participants
  Week 6: number analyzed (Participants) | 22 | 12
  Week 6 | 8 | 2
  Week 12: number analyzed (Participants) | 13 | 5
  Week 12 | 7 | 1
  Month 9: number analyzed (Participants) | 11 | 4
  Month 9 | 0 | 1
  Month 18: number analyzed (Participants) | 7 | 4
  Month 18 | 2 | 0
  Month 24: number analyzed (Participants) | 10 | 4
  Month 24 | 1 | 1
  Month 30: number analyzed (Participants) | 5 | 2
  Month 30 | 2 | 1
  FU visit: number analyzed (Participants) | 10 | 3
  FU visit | 2 | 0
  Any | 15 | 1

10. Secondary Outcome: Number of Subjects With Cell-mediated Immunity (CMI) Cluster of Differentiation (CD) 8+ Response
Description: Responders were patients with at least 5x10-⁶ increase in minimal CD8 precursor frequency versus baseline. Any = at least one post treatment time point.
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 34 | 16
Participants
  Week 6: number analyzed (Participants) | 19 | 11
  Week 6 | 2 | 3
  Week 12: number analyzed (Participants) | 10 | 7
  Week 12 | 1 | 0
  Month 9: number analyzed (Participants) | 12 | 5
  Month 9 | 3 | 1
  Month 18: number analyzed (Participants) | 8 | 3
  Month 18 | 3 | 1
  Month 24: number analyzed (Participants) | 10 | 5
  Month 24 | 0 | 1
  Month 30: number analyzed (Participants) | 7 | 0
  Month 30 | 1 | 0
  FU visit: number analyzed (Participants) | 9 | 3
  FU visit | 1 | 1
  Any | 9 | 6

11. Secondary Outcome: Number of Subjects With Cell-mediated Immunity (CMI) CD4+ or CD8+ Response
Description: Responders are patients with at least 5x10-⁶ increase in minimal CD4 or CD8 precursor frequency versus baseline. Any = at least one post treatment time point.
Time Frame: At Week 6, Week 12, Month 9, Month 18, Month 24, at Month 30 and at Month 60
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 40 | 18
Participants
  Week 6: number analyzed (Participants) | 24 | 13
  Week 6 | 10 | 5
  Week 12: number analyzed (Participants) | 15 | 7
  Week 12 | 8 | 1
  Month 9: number analyzed (Participants) | 13 | 5
  Month 9 | 3 | 2
  Month 18: number analyzed (Participants) | 8 | 4
  Month 18 | 3 | 1
  Month 24: number analyzed (Participants) | 11 | 6
  Month 24 | 1 | 1
  Month 30: number analyzed (Participants) | 7 | 2
  Month 30 | 2 | 1
  Month 60: number analyzed (Participants) | 10 | 3
  Month 60 | 2 | 1
  Any | 21 | 7

12. Secondary Outcome: Number of Patients Reporting Non-small-cell Lung Cancer (NSCLC) Recurrence by Gene Signature
Description: Types of recurrence included local, regional and distant metastasis and second primary lung tumours, and comprised: Local recurrence, defined as a tumour within the same lung or at the bronchial stump; Regional recurrence, involving a clinically or radiologically manifest disease in the mediastinum or in supraclavicular nodes; and Distant recurrence, i.e., any tumour arising in the contralateral lung or outside the hemithorax. Gene expression profiling was performed by qRT-PCR in primary tumor samples taken at the time of resection of the tumor, and thus before any study treatment. Gene signature positive (GS+) and negative (GS-) profiles were assessed with a 61-set gene signature (GS) and a classifier which were defined in the Phase II melanoma EORTC 16032-18031 study.
Time Frame: Over a median follow up time of 86 months
Population: Analysis was performed on the Total Treated cohort Gene Signature set which included all subjects of the Total Treated cohort for whom ribonucleic acid (RNA) from their tumour samples was available to perform the gene signature test.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 106 | 51
Participants
  GS+: number analyzed (Participants) | 41 | 20
  GS+ | 13 | 9
  GS-: number analyzed (Participants) | 65 | 31
  GS- | 31 | 12

13. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 8-day (Days 0-7) post-vaccination period, across doses
Population: The analyses were performed on the Total Treated cohort, which included all patients who were randomised and who received at least one dose of the randomised study product administration and with a documented symptom sheet.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 121 | 58
Participants
  Any Pain | 116 | 36
  Grade 3 Pain | 59 | 2
  Any Redness | 96 | 24
  Grade 3 Redness | 66 | 2
  Any Swelling | 91 | 19
  Grade 3 Swelling | 52 | 4

14. Secondary Outcome: Number of Subjects With Any, Grade 2/3/4 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, headache, myalgia, nasea, rigors/chills, sweating/diaphoresis, temperature [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], vomiting. Any = occurrence of the symptom regardless of intensity grade. Grade 4 Fatigue = Bedridden or disabling. Grade 4 Headache, Myalgia = Disabling. Grade 3 Nausea = No significant intake, requiring i.v. fluids. Grade 3 Rigors/Chills = Not responsive to narcotic medication. Grade 2 Sweating/Diaphoresis = Frequent or drenching. Grade 4 Vomiting = Requiring parenteral nutrition; or physiologic consequences requiring intensive care; haemodynamic collapse. Grade 3 fever = fever higher than (>) 40.0 °C for more than 24 hours. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 8-day (Days 0-7) post-vaccination period, across doses
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 121 | 58
Participants
  Any Fatigue | 87 | 32
  Grade 4 Fatigue | 2 | 1
  Related Fatigue | 78 | 23
  Any Headache | 81 | 24
  Grade 4 Headache | 1 | 0
  Related Headache | 69 | 16
  Any Myalgia | 90 | 29
  Grade 4 Myalgia | 5 | 1
  Related Myalgia | 77 | 24
  Any Nausea | 46 | 18
  Grade 3 Nausea | 1 | 0
  Related Nausea | 42 | 15
  Any Rigors/Chills | 62 | 13
  Grade 3 Rigors/Chills | 8 | 0
  Any Sweating/Diaphoresis | 62 | 19
  Grade 2 Sweating/Diaphoresis | 25 | 9
  Related Sweating/Diaphoresis | 53 | 16
  Any Temperature | 45 | 8
  Grade 3 Temperature | 0 | 0
  Related Temperature | 40 | 3
  Any Vomiting | 16 | 9
  Grade 4 Vomiting | 0 | 0
  Related Vomiting | 13 | 7

15. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within the 31-day (Days 0-30) post-vaccination period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 122 | 60
Participants | 95 | 50

16. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout the study (Day 0 - Month 86)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 122 | 60
Participants | 41 | 21

17. Secondary Outcome: Number of Subjects With Normal and Abnormal Urinalysis Parameters
Description: The parameters analysed were Protein, Red Blood Cells (RBC) and White Blood Cells (WBC), with respect to normal laboratory ranges. The subjects were grouped by status at baseline.
Time Frame: At Month 6, Month 12, Month 18, Month 24 and Month 30
Population: The analyses were performed on the Total Treated cohort gene signature (GS) set, which included all subjects of the Total Treated cohort for whom ribonucleic acid (RNA) from their tumour samples was available to perform the gene signature test and with data available for the considered assay.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 100 | 50
Participants
  Protein, Normal values at Baseline, Month 6: Normal | 100 | 50
  Protein, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  Protein, Normal values at Baseline, Month 12: number analyzed (Participants) | 86 | 38
  Protein, Normal values at Baseline, Month 12: Normal | 86 | 38
  Protein, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  Protein, Normal values at Baseline, Month 18: number analyzed (Participants) | 72 | 33
  Protein, Normal values at Baseline, Month 18: Normal | 72 | 33
  Protein, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  Protein, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  Protein, Normal values at Baseline, Month 24: Normal | 68 | 31
  Protein, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  Protein, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 23
  Protein, Normal values at Baseline, Month 30: Normal | 55 | 23
  Protein, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  RBC, Normal values at Baseline, Month 6: Normal | 100 | 50
  RBC, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  RBC, Normal values at Baseline, Month 12: number analyzed (Participants) | 86 | 38
  RBC, Normal values at Baseline, Month 12: Normal | 86 | 38
  RBC, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  RBC, Normal values at Baseline, Month 18: number analyzed (Participants) | 72 | 33
  RBC, Normal values at Baseline, Month 18: Normal | 72 | 33
  RBC, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  RBC, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  RBC, Normal values at Baseline, Month 24: Normal | 68 | 31
  RBC, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  RBC, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 23
  RBC, Normal values at Baseline, Month 30: Normal | 55 | 23
  RBC, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  WBC, Normal values at Baseline, Month 6: Normal | 100 | 50
  WBC, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  WBC, Normal values at Baseline, Month 12: number analyzed (Participants) | 86 | 38
  WBC, Normal values at Baseline, Month 12: Normal | 86 | 38
  WBC, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  WBC, Normal values at Baseline, Month 18: number analyzed (Participants) | 72 | 33
  WBC, Normal values at Baseline, Month 18: Normal | 72 | 33
  WBC, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  WBC, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  WBC, Normal values at Baseline, Month 24: Normal | 68 | 31
  WBC, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  WBC, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 23
  WBC, Normal values at Baseline, Month 30: Normal | 55 | 23
  WBC, Normal values at Baseline, Month 30: Abnormal | 0 | 0

18. Secondary Outcome: Number of Subjects With Normal and Abnormal Hematological Parameters
Description: The parameters analysed were Basophils (BAS), Eosinophils (EOS), Haemoglobin (HGB), Lymphocytes (LYM), Monocytes (MON), Neutrophils (NEU), Platelets (PLA), Red Blood Cells (RBC), Sedimentations rate (SED) and White Blood Cells (WBC), with respect to normal laboratory ranges. The subjects were grouped by status at baseline.
Time Frame: At Month 6, Month 12, Month 18, Month 24 and Month 30
Population: The analyses were performed on the Total Treated cohort, which included all patients who were randomised and who received at least one dose of the randomised study product administration and with data available for the respective assay.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 122 | 59
Participants
  BAS, Normal values at Baseline, Month 6: Normal | 122 | 59
  BAS, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  BAS, Normal values at Baseline, Month 12: number analyzed (Participants) | 121 | 59
  BAS, Normal values at Baseline, Month 12: Normal | 121 | 59
  BAS, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  BAS, Normal values at Baseline, Month 18: Normal | 122 | 59
  BAS, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  BAS, Normal values at Baseline, Month 24: number analyzed (Participants) | 120 | 59
  BAS, Normal values at Baseline, Month 24: Normal | 120 | 59
  BAS, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  BAS, Normal values at Baseline, Month 30: number analyzed (Participants) | 111 | 51
  BAS, Normal values at Baseline, Month 30: Normal | 111 | 51
  BAS, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  EOS, Normal values at Baseline, Month 6: Normal | 122 | 59
  EOS, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  EOS, Normal values at Baseline, Month 12: number analyzed (Participants) | 121 | 59
  EOS, Normal values at Baseline, Month 12: Normal | 121 | 59
  EOS, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  EOS, Normal values at Baseline, Month 18: Normal | 122 | 59
  EOS, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  EOS, Normal values at Baseline, Month 24: number analyzed (Participants) | 120 | 59
  EOS, Normal values at Baseline, Month 24: Normal | 120 | 59
  EOS, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  EOS, Normal values at Baseline, Month 30: number analyzed (Participants) | 111 | 51
  EOS, Normal values at Baseline, Month 30: Normal | 111 | 51
  EOS, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  HGB, Normal values at Baseline, Month 6: Normal | 122 | 59
  HGB, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  HGB, Normal values at Baseline, Month 12: number analyzed (Participants) | 121 | 59
  HGB, Normal values at Baseline, Month 12: Normal | 121 | 59
  HGB, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  HGB, Normal values at Baseline, Month 18: Normal | 122 | 59
  HGB, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  HGB, Normal values at Baseline, Month 24: number analyzed (Participants) | 120 | 59
  HGB, Normal values at Baseline, Month 24: Normal | 120 | 59
  HGB, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  HGB, Normal values at Baseline, Month 30: number analyzed (Participants) | 111 | 51
  HGB, Normal values at Baseline, Month 30: Normal | 111 | 51
  HGB, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  LYM, Normal values at Baseline, Month 6: number analyzed (Participants) | 121 | 59
  LYM, Normal values at Baseline, Month 6: Normal | 121 | 59
  LYM, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  LYM, Normal values at Baseline, Month 12: number analyzed (Participants) | 120 | 59
  LYM, Normal values at Baseline, Month 12: Normal | 120 | 59
  LYM, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  LYM, Normal values at Baseline, Month 18: number analyzed (Participants) | 121 | 59
  LYM, Normal values at Baseline, Month 18: Normal | 121 | 59
  LYM, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  LYM, Normal values at Baseline, Month 24: number analyzed (Participants) | 119 | 59
  LYM, Normal values at Baseline, Month 24: Normal | 119 | 59
  LYM, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  LYM, Normal values at Baseline, Month 30: number analyzed (Participants) | 110 | 51
  LYM, Normal values at Baseline, Month 30: Normal | 109 | 51
  LYM, Normal values at Baseline, Month 30: Abnormal | 1 | 0
  LYM, Abnormal values at Baseline, Month 6: number analyzed (Participants) | 1 | 0
  LYM, Abnormal values at Baseline, Month 6: Normal | 1 | 0
  LYM, Abnormal values at Baseline, Month 6: Abnormal | 0 | 0
  LYM, Abnormal values at Baseline, Month 12: number analyzed (Participants) | 1 | 0
  LYM, Abnormal values at Baseline, Month 12: Normal | 1 | 0
  LYM, Abnormal values at Baseline, Month 12: Abnormal | 0 | 0
  LYM, Abnormal values at Baseline, Month 18: number analyzed (Participants) | 1 | 0
  LYM, Abnormal values at Baseline, Month 18: Normal | 1 | 0
  LYM, Abnormal values at Baseline, Month 18: Abnormal | 0 | 0
  LYM, Abnormal values at Baseline, Month 24: number analyzed (Participants) | 1 | 0
  LYM, Abnormal values at Baseline, Month 24: Normal | 1 | 0
  LYM, Abnormal values at Baseline, Month 24: Abnormal | 0 | 0
  LYM, Abnormal values at Baseline, Month 30: number analyzed (Participants) | 1 | 0
  LYM, Abnormal values at Baseline, Month 30: Normal | 1 | 0
  LYM, Abnormal values at Baseline, Month 30: Abnormal | 0 | 0
  MON, Normal values at Baseline, Month 6: Normal | 122 | 59
  MON, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  MON, Normal values at Baseline, Month 12: number analyzed (Participants) | 121 | 59
  MON, Normal values at Baseline, Month 12: Normal | 121 | 59
  MON, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  MON, Normal values at Baseline, Month 18: Normal | 122 | 59
  MON, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  MON, Normal values at Baseline, Month 24: number analyzed (Participants) | 120 | 59
  MON, Normal values at Baseline, Month 24: Normal | 120 | 59
  MON, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  MON, Normal values at Baseline, Month 30: number analyzed (Participants) | 111 | 51
  MON, Normal values at Baseline, Month 30: Normal | 111 | 51
  MON, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  NEU, Normal values at Baseline, Month 6: Normal | 122 | 59
  NEU, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  NEU, Normal values at Baseline, Month 12: number analyzed (Participants) | 121 | 59
  NEU, Normal values at Baseline, Month 12: Normal | 121 | 59
  NEU, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  NEU, Normal values at Baseline, Month 18: Normal | 122 | 59
  NEU, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  NEU, Normal values at Baseline, Month 24: number analyzed (Participants) | 120 | 59
  NEU, Normal values at Baseline, Month 24: Normal | 120 | 59
  NEU, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  NEU, Normal values at Baseline, Month 30: number analyzed (Participants) | 111 | 51
  NEU, Normal values at Baseline, Month 30: Normal | 110 | 51
  NEU, Normal values at Baseline, Month 30: Abnormal | 1 | 0
  PLA, Normal values at Baseline, Month 6: Normal | 122 | 59
  PLA, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  PLA, Normal values at Baseline, Month 12: number analyzed (Participants) | 121 | 59
  PLA, Normal values at Baseline, Month 12: Normal | 121 | 59
  PLA, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  PLA, Normal values at Baseline, Month 18: Normal | 122 | 59
  PLA, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  PLA, Normal values at Baseline, Month 24: number analyzed (Participants) | 120 | 59
  PLA, Normal values at Baseline, Month 24: Normal | 120 | 59
  PLA, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  PLA, Normal values at Baseline, Month 30: number analyzed (Participants) | 111 | 51
  PLA, Normal values at Baseline, Month 30: Normal | 111 | 51
  PLA, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  RBC, Normal values at Baseline, Month 6: Normal | 122 | 59
  RBC, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  RBC, Normal values at Baseline, Month 12: number analyzed (Participants) | 121 | 59
  RBC, Normal values at Baseline, Month 12: Normal | 121 | 59
  RBC, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  RBC, Normal values at Baseline, Month 18: Normal | 122 | 59
  RBC, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  RBC, Normal values at Baseline, Month 24: number analyzed (Participants) | 120 | 59
  RBC, Normal values at Baseline, Month 24: Normal | 120 | 59
  RBC, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  RBC, Normal values at Baseline, Month 30: number analyzed (Participants) | 111 | 51
  RBC, Normal values at Baseline, Month 30: Normal | 111 | 51
  RBC, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  SED, Normal values at Baseline, Month 6: Normal | 122 | 59
  SED, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  SED, Normal values at Baseline, Month 12: number analyzed (Participants) | 121 | 59
  SED, Normal values at Baseline, Month 12: Normal | 121 | 59
  SED, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  SED, Normal values at Baseline, Month 18: Normal | 122 | 59
  SED, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  SED, Normal values at Baseline, Month 24: number analyzed (Participants) | 120 | 59
  SED, Normal values at Baseline, Month 24: Normal | 120 | 59
  SED, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  SED, Normal values at Baseline, Month 30: number analyzed (Participants) | 111 | 51
  SED, Normal values at Baseline, Month 30: Normal | 111 | 51
  SED, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  WBC, Normal values at Baseline, Month 6: Normal | 122 | 59
  WBC, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  WBC, Normal values at Baseline, Month 12: number analyzed (Participants) | 121 | 59
  WBC, Normal values at Baseline, Month 12: Normal | 121 | 59
  WBC, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  WBC, Normal values at Baseline, Month 18: Normal | 122 | 59
  WBC, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  WBC, Normal values at Baseline, Month 24: number analyzed (Participants) | 120 | 59
  WBC, Normal values at Baseline, Month 24: Normal | 120 | 59
  WBC, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  WBC, Normal values at Baseline, Month 30: number analyzed (Participants) | 111 | 51
  WBC, Normal values at Baseline, Month 30: Normal | 110 | 51
  WBC, Normal values at Baseline, Month 30: Abnormal | 1 | 0

19. Secondary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters
Description: The parameters analysed were Albumin (ALB), Bicarbonate (BIC), Blood urea nitrogen (BUN), Calcium (CAL), Chloride (CHL), Cholesterol (CHO), Creatinine (CREA), Glucose (GLU), Magnesium (MAG), Phosphate (PHO), Potassium (POT), Sodium (SOD), Total protein (TPROT), Total bilirubin (TBIL), Triglycerides (TRIG) and Uric acid (UAC), with respect to normal laboratory ranges. The subjects were grouped by status at baseline.
Time Frame: At Month 6, Month 12, Month 18, Month 24 and Month 30
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 249553 Group | Placebo Group
Number analyzed (Participants) | 97 | 45
Participants
  ALB, Normal values at Baseline, Month 6: Normal | 97 | 45
  ALB, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  ALB, Normal values at Baseline, Month 12: number analyzed (Participants) | 85 | 34
  ALB, Normal values at Baseline, Month 12: Normal | 85 | 33
  ALB, Normal values at Baseline, Month 12: Abnormal | 0 | 1
  ALB, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 30
  ALB, Normal values at Baseline, Month 18: Normal | 70 | 30
  ALB, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  ALB, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  ALB, Normal values at Baseline, Month 24: Normal | 68 | 31
  ALB, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  ALB, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 22
  ALB, Normal values at Baseline, Month 30: Normal | 55 | 22
  ALB, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  BIC, Normal values at Baseline, Month 6: Normal | 97 | 45
  BIC, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  BIC, Normal values at Baseline, Month 12: number analyzed (Participants) | 85 | 34
  BIC, Normal values at Baseline, Month 12: Normal | 85 | 34
  BIC, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  BIC, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 30
  BIC, Normal values at Baseline, Month 18: Normal | 70 | 30
  BIC, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  BIC, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  BIC, Normal values at Baseline, Month 24: Normal | 68 | 31
  BIC, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  BIC, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 22
  BIC, Normal values at Baseline, Month 30: Normal | 55 | 22
  BIC, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  BUN, Normal values at Baseline, Month 6: Normal | 97 | 45
  BUN, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  BUN, Normal values at Baseline, Month 12: number analyzed (Participants) | 85 | 34
  BUN, Normal values at Baseline, Month 12: Normal | 85 | 34
  BUN, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  BUN, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 30
  BUN, Normal values at Baseline, Month 18: Normal | 70 | 30
  BUN, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  BUN, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  BUN, Normal values at Baseline, Month 24: Normal | 68 | 31
  BUN, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  BUN, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 22
  BUN, Normal values at Baseline, Month 30: Normal | 55 | 22
  BUN, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  CAL, Normal values at Baseline, Month 6: number analyzed (Participants) | 92 | 44
  CAL, Normal values at Baseline, Month 6: Normal | 91 | 43
  CAL, Normal values at Baseline, Month 6: Abnormal | 1 | 1
  CAL, Normal values at Baseline, Month 12: number analyzed (Participants) | 80 | 34
  CAL, Normal values at Baseline, Month 12: Normal | 80 | 33
  CAL, Normal values at Baseline, Month 12: Abnormal | 0 | 1
  CAL, Normal values at Baseline, Month 18: number analyzed (Participants) | 67 | 30
  CAL, Normal values at Baseline, Month 18: Normal | 67 | 30
  CAL, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  CAL, Normal values at Baseline, Month 24: number analyzed (Participants) | 65 | 31
  CAL, Normal values at Baseline, Month 24: Normal | 65 | 30
  CAL, Normal values at Baseline, Month 24: Abnormal | 0 | 1
  CAL, Normal values at Baseline, Month 30: number analyzed (Participants) | 53 | 22
  CAL, Normal values at Baseline, Month 30: Normal | 53 | 22
  CAL, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  CAL, Abnormal values at Baseline, Month 6: number analyzed (Participants) | 5 | 1
  CAL, Abnormal values at Baseline, Month 6: Normal | 2 | 0
  CAL, Abnormal values at Baseline, Month 6: Abnormal | 3 | 1
  CAL, Abnormal values at Baseline, Month 12: number analyzed (Participants) | 5 | 0
  CAL, Abnormal values at Baseline, Month 12: Normal | 2 | 0
  CAL, Abnormal values at Baseline, Month 12: Abnormal | 3 | 0
  CAL, Abnormal values at Baseline, Month 18: number analyzed (Participants) | 3 | 0
  CAL, Abnormal values at Baseline, Month 18: Normal | 1 | 0
  CAL, Abnormal values at Baseline, Month 18: Abnormal | 2 | 0
  CAL, Abnormal values at Baseline, Month 24: number analyzed (Participants) | 3 | 0
  CAL, Abnormal values at Baseline, Month 24: Normal | 1 | 0
  CAL, Abnormal values at Baseline, Month 24: Abnormal | 2 | 0
  CAL, Abnormal values at Baseline, Month 30: number analyzed (Participants) | 2 | 0
  CAL, Abnormal values at Baseline, Month 30: Normal | 2 | 0
  CAL, Abnormal values at Baseline, Month 30: Abnormal | 0 | 0
  CHL, Normal values at Baseline, Month 6: Normal | 97 | 45
  CHL, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  CHL, Normal values at Baseline, Month 12: number analyzed (Participants) | 85 | 34
  CHL, Normal values at Baseline, Month 12: Normal | 85 | 34
  CHL, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  CHL, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 30
  CHL, Normal values at Baseline, Month 18: Normal | 70 | 30
  CHL, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  CHL, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  CHL, Normal values at Baseline, Month 24: Normal | 68 | 31
  CHL, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  CHL, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 22
  CHL, Normal values at Baseline, Month 30: Normal | 55 | 22
  CHL, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  CHO, Normal values at Baseline, Month 6: number analyzed (Participants) | 97 | 44
  CHO, Normal values at Baseline, Month 6: Normal | 96 | 44
  CHO, Normal values at Baseline, Month 6: Abnormal | 1 | 0
  CHO, Normal values at Baseline, Month 12: number analyzed (Participants) | 85 | 33
  CHO, Normal values at Baseline, Month 12: Normal | 85 | 33
  CHO, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  CHO, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 29
  CHO, Normal values at Baseline, Month 18: Normal | 70 | 29
  CHO, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  CHO, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 30
  CHO, Normal values at Baseline, Month 24: Normal | 68 | 30
  CHO, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  CHO, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 21
  CHO, Normal values at Baseline, Month 30: Normal | 55 | 21
  CHO, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  CHO, Abnormal values at Baseline, Month 6: number analyzed (Participants) | 0 | 1
  CHO, Abnormal values at Baseline, Month 6: Normal | 0 | 1
  CHO, Abnormal values at Baseline, Month 6: Abnormal | 0 | 0
  CHO, Abnormal values at Baseline, Month 12: number analyzed (Participants) | 0 | 1
  CHO, Abnormal values at Baseline, Month 12: Normal | 0 | 1
  CHO, Abnormal values at Baseline, Month 12: Abnormal | 0 | 0
  CHO, Abnormal values at Baseline, Month 18: number analyzed (Participants) | 0 | 1
  CHO, Abnormal values at Baseline, Month 18: Normal | 0 | 1
  CHO, Abnormal values at Baseline, Month 18: Abnormal | 0 | 0
  CHO, Abnormal values at Baseline, Month 24: number analyzed (Participants) | 0 | 1
  CHO, Abnormal values at Baseline, Month 24: Normal | 0 | 1
  CHO, Abnormal values at Baseline, Month 24: Abnormal | 0 | 0
  CHO, Abnormal values at Baseline, Month 30: number analyzed (Participants) | 0 | 1
  CHO, Abnormal values at Baseline, Month 30: Normal | 0 | 1
  CHO, Abnormal values at Baseline, Month 30: Abnormal | 0 | 0
  CREA, Normal values at Baseline, Month 6: Normal | 97 | 45
  CREA, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  CREA, Normal values at Baseline, Month 12: number analyzed (Participants) | 85 | 34
  CREA, Normal values at Baseline, Month 12: Normal | 84 | 34
  CREA, Normal values at Baseline, Month 12: Abnormal | 1 | 0
  CREA, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 30
  CREA, Normal values at Baseline, Month 18: Normal | 69 | 30
  CREA, Normal values at Baseline, Month 18: Abnormal | 1 | 0
  CREA, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  CREA, Normal values at Baseline, Month 24: Normal | 68 | 31
  CREA, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  CREA, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 22
  CREA, Normal values at Baseline, Month 30: Normal | 55 | 22
  CREA, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  GLU, Normal values at Baseline, Month 6: number analyzed (Participants) | 96 | 45
  GLU, Normal values at Baseline, Month 6: Normal | 94 | 45
  GLU, Normal values at Baseline, Month 6: Abnormal | 2 | 0
  GLU, Normal values at Baseline, Month 12: number analyzed (Participants) | 84 | 33
  GLU, Normal values at Baseline, Month 12: Normal | 83 | 32
  GLU, Normal values at Baseline, Month 12: Abnormal | 1 | 1
  GLU, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 29
  GLU, Normal values at Baseline, Month 18: Normal | 70 | 28
  GLU, Normal values at Baseline, Month 18: Abnormal | 0 | 1
  GLU, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 30
  GLU, Normal values at Baseline, Month 24: Normal | 67 | 29
  GLU, Normal values at Baseline, Month 24: Abnormal | 1 | 1
  GLU, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 22
  GLU, Normal values at Baseline, Month 30: Normal | 54 | 22
  GLU, Normal values at Baseline, Month 30: Abnormal | 1 | 0
  GLU, Abnormal values at Baseline, Month 6: number analyzed (Participants) | 1 | 0
  GLU, Abnormal values at Baseline, Month 6: Normal | 1 | 0
  GLU, Abnormal values at Baseline, Month 6: Abnormal | 0 | 0
  GLU, Abnormal values at Baseline, Month 12: number analyzed (Participants) | 1 | 1
  GLU, Abnormal values at Baseline, Month 12: Normal | 1 | 1
  GLU, Abnormal values at Baseline, Month 12: Abnormal | 0 | 0
  GLU, Abnormal values at Baseline, Month 18: number analyzed (Participants) | 0 | 1
  GLU, Abnormal values at Baseline, Month 18: Normal | 0 | 1
  GLU, Abnormal values at Baseline, Month 18: Abnormal | 0 | 0
  GLU, Abnormal values at Baseline, Month 24: number analyzed (Participants) | 0 | 1
  GLU, Abnormal values at Baseline, Month 24: Normal | 0 | 1
  GLU, Abnormal values at Baseline, Month 24: Abnormal | 0 | 0
  MAG, Normal values at Baseline, Month 6: number analyzed (Participants) | 96 | 45
  MAG, Normal values at Baseline, Month 6: Normal | 96 | 45
  MAG, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  MAG, Normal values at Baseline, Month 12: number analyzed (Participants) | 84 | 34
  MAG, Normal values at Baseline, Month 12: Normal | 83 | 34
  MAG, Normal values at Baseline, Month 12: Abnormal | 1 | 0
  MAG, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 30
  MAG, Normal values at Baseline, Month 18: Normal | 70 | 30
  MAG, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  MAG, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  MAG, Normal values at Baseline, Month 24: Normal | 68 | 30
  MAG, Normal values at Baseline, Month 24: Abnormal | 0 | 1
  MAG, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 22
  MAG, Normal values at Baseline, Month 30: Normal | 55 | 22
  MAG, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  MAG, Abnormal values at Baseline, Month 6: number analyzed (Participants) | 1 | 0
  MAG, Abnormal values at Baseline, Month 6: Normal | 1 | 0
  MAG, Abnormal values at Baseline, Month 6: Abnormal | 0 | 0
  MAG, Abnormal values at Baseline, Month 12: number analyzed (Participants) | 1 | 0
  MAG, Abnormal values at Baseline, Month 12: Normal | 1 | 0
  MAG, Abnormal values at Baseline, Month 12: Abnormal | 0 | 0
  PHO, Normal values at Baseline, Month 6: Normal | 97 | 45
  PHO, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  PHO, Normal values at Baseline, Month 12: number analyzed (Participants) | 85 | 34
  PHO, Normal values at Baseline, Month 12: Normal | 85 | 34
  PHO, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  PHO, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 30
  PHO, Normal values at Baseline, Month 18: Normal | 70 | 30
  PHO, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  PHO, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  PHO, Normal values at Baseline, Month 24: Normal | 68 | 31
  PHO, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  PHO, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 22
  PHO, Normal values at Baseline, Month 30: Normal | 55 | 22
  PHO, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  POT, Normal values at Baseline, Month 6: Normal | 96 | 45
  POT, Normal values at Baseline, Month 6: Abnormal | 1 | 0
  POT, Normal values at Baseline, Month 12: number analyzed (Participants) | 85 | 34
  POT, Normal values at Baseline, Month 12: Normal | 85 | 34
  POT, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  POT, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 30
  POT, Normal values at Baseline, Month 18: Normal | 70 | 30
  POT, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  POT, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  POT, Normal values at Baseline, Month 24: Normal | 68 | 31
  POT, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  POT, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 22
  POT, Normal values at Baseline, Month 30: Normal | 55 | 22
  POT, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  SOD, Normal values at Baseline, Month 6: Normal | 97 | 45
  SOD, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  SOD, Normal values at Baseline, Month 12: number analyzed (Participants) | 85 | 34
  SOD, Normal values at Baseline, Month 12: Normal | 85 | 34
  SOD, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  SOD, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 30
  SOD, Normal values at Baseline, Month 18: Normal | 70 | 30
  SOD, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  SOD, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  SOD, Normal values at Baseline, Month 24: Normal | 67 | 31
  SOD, Normal values at Baseline, Month 24: Abnormal | 1 | 0
  SOD, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 22
  SOD, Normal values at Baseline, Month 30: Normal | 55 | 22
  SOD, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  TPROT, Normal values at Baseline, Month 6: Normal | 97 | 45
  TPROT, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  TPROT, Normal values at Baseline, Month 12: number analyzed (Participants) | 85 | 34
  TPROT, Normal values at Baseline, Month 12: Normal | 85 | 34
  TPROT, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  TPROT, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 30
  TPROT, Normal values at Baseline, Month 18: Normal | 70 | 30
  TPROT, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  TPROT, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  TPROT, Normal values at Baseline, Month 24: Normal | 68 | 31
  TPROT, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  TPROT, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 22
  TPROT, Normal values at Baseline, Month 30: Normal | 55 | 22
  TPROT, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  TBIL, Normal values at Baseline, Month 6: Normal | 97 | 45
  TBIL, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  TBIL, Normal values at Baseline, Month 12: number analyzed (Participants) | 85 | 34
  TBIL, Normal values at Baseline, Month 12: Normal | 85 | 34
  TBIL, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  TBIL, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 30
  TBIL, Normal values at Baseline, Month 18: Normal | 70 | 30
  TBIL, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  TBIL, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  TBIL, Normal values at Baseline, Month 24: Normal | 68 | 31
  TBIL, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  TBIL, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 22
  TBIL, Normal values at Baseline, Month 30: Normal | 55 | 22
  TBIL, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  TRIG, Normal values at Baseline, Month 6: number analyzed (Participants) | 97 | 44
  TRIG, Normal values at Baseline, Month 6: Normal | 97 | 44
  TRIG, Normal values at Baseline, Month 6: Abnormal | 0 | 0
  TRIG, Normal values at Baseline, Month 12: number analyzed (Participants) | 85 | 33
  TRIG, Normal values at Baseline, Month 12: Normal | 85 | 33
  TRIG, Normal values at Baseline, Month 12: Abnormal | 0 | 0
  TRIG, Normal values at Baseline, Month 18: number analyzed (Participants) | 70 | 29
  TRIG, Normal values at Baseline, Month 18: Normal | 70 | 29
  TRIG, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  TRIG, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 30
  TRIG, Normal values at Baseline, Month 24: Normal | 68 | 30
  TRIG, Normal values at Baseline, Month 24: Abnormal | 0 | 0
  TRIG, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 21
  TRIG, Normal values at Baseline, Month 30: Normal | 55 | 21
  TRIG, Normal values at Baseline, Month 30: Abnormal | 0 | 0
  TRIG, Abnormal values at Baseline, Month 6: number analyzed (Participants) | 0 | 1
  TRIG, Abnormal values at Baseline, Month 6: Normal | 0 | 1
  TRIG, Abnormal values at Baseline, Month 6: Abnormal | 0 | 0
  TRIG, Abnormal values at Baseline, Month 12: number analyzed (Participants) | 0 | 1
  TRIG, Abnormal values at Baseline, Month 12: Normal | 0 | 1
  TRIG, Abnormal values at Baseline, Month 12: Abnormal | 0 | 0
  TRIG, Abnormal values at Baseline, Month 18: number analyzed (Participants) | 0 | 1
  TRIG, Abnormal values at Baseline, Month 18: Normal | 0 | 1
  TRIG, Abnormal values at Baseline, Month 18: Abnormal | 0 | 0
  TRIG, Abnormal values at Baseline, Month 24: number analyzed (Participants) | 0 | 1
  TRIG, Abnormal values at Baseline, Month 24: Normal | 0 | 1
  TRIG, Abnormal values at Baseline, Month 24: Abnormal | 0 | 0
  TRIG, Abnormal values at Baseline, Month 30: number analyzed (Participants) | 0 | 1
  TRIG, Abnormal values at Baseline, Month 30: Normal | 0 | 1
  TRIG, Abnormal values at Baseline, Month 30: Abnormal | 0 | 0
  UAC, Normal values at Baseline, Month 6: number analyzed (Participants) | 96 | 45
  UAC, Normal values at Baseline, Month 6: Normal | 95 | 44
  UAC, Normal values at Baseline, Month 6: Abnormal | 1 | 1
  UAC, Normal values at Baseline, Month 12: number analyzed (Participants) | 84 | 34
  UAC, Normal values at Baseline, Month 12: Normal | 83 | 34
  UAC, Normal values at Baseline, Month 12: Abnormal | 1 | 0
  UAC, Normal values at Baseline, Month 18: number analyzed (Participants) | 69 | 30
  UAC, Normal values at Baseline, Month 18: Normal | 69 | 30
  UAC, Normal values at Baseline, Month 18: Abnormal | 0 | 0
  UAC, Normal values at Baseline, Month 24: number analyzed (Participants) | 68 | 31
  UAC, Normal values at Baseline, Month 24: Normal | 68 | 29
  UAC, Normal values at Baseline, Month 24: Abnormal | 0 | 2
  UAC, Normal values at Baseline, Month 30: number analyzed (Participants) | 55 | 22
  UAC, Normal values at Baseline, Month 30: Normal | 54 | 22
  UAC, Normal values at Baseline, Month 30: Abnormal | 1 | 0
  UAC, Abnormal values at Baseline, Month 6: number analyzed (Participants) | 1 | 0
  UAC, Abnormal values at Baseline, Month 6: Normal | 1 | 0
  UAC, Abnormal values at Baseline, Month 6: Abnormal | 0 | 0
  UAC, Abnormal values at Baseline, Month 12: number analyzed (Participants) | 1 | 0
  UAC, Abnormal values at Baseline, Month 12: Normal | 1 | 0
  UAC, Abnormal values at Baseline, Month 12: Abnormal | 0 | 0
  UAC, Abnormal values at Baseline, Month 18: number analyzed (Participants) | 1 | 0
  UAC, Abnormal values at Baseline, Month 18: Normal | 1 | 0
  UAC, Abnormal values at Baseline, Month 18: Abnormal | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and SAEs: during the entire study period (Month 0 up to Month 86). Other Adverse Events - Solicited local and general symptoms: during the 8-day (Days 0-7) post-product administration period; - Unsolicited AEs: within the 31-day (Days 0-30) post-product administration period.
Description: Deaths, as study events, were not all recorded as SAEs. Only deaths occurring in patients without recurrence during the Treatment Phase of the study (up to Month 30) and recorded as fatal SAEs are reported and not all deaths reported without recurrence were classified as fatal SAEs.
Arm/Group | GSK 249553 Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 54/122 | 26/60
Serious Adverse Events (participants affected / at risk) | 41/122 | 21/60
Other Adverse Events (participants affected / at risk) | 120/122 | 53/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK 249553 Group (N=122) | Placebo Group (N=60)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Inguinal hernia (Musculoskeletal and connective tissue disorders) | 1 | 1
Adrenal gland cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial fistula (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cerebral ischemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colonic polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic foot (Infections and infestations) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Empyema (Infections and infestations) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastritis (Metabolism and nutrition disorders) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hyperglycaemia (Blood and lymphatic system disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Lymphocele (Blood and lymphatic system disorders) | 1 | 0
Malaise (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myocardial ischemia (Cardiac disorders) | 0 | 1
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatitis acute (Infections and infestations) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Peripheral ischemia (Nervous system disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Infections and infestations) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 1 | 0
Sciatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Small cell lung cancer stage unspecified (Skin and subcutaneous tissue disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Syncope (Vascular disorders) | 1 | 0
Thoracic outlet syndrome (Vascular disorders) | 1 | 0
Urethral cancer (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Bladder transitional cell carcinoma (Renal and urinary disorders) | 1 | 0
Metastases to kidney (Renal and urinary disorders) | 1 | 0
Medical observation (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK 249553 Group (N=122) | Placebo Group (N=60)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Bronchitis (Infections and infestations) | 7 (10) | 0 (0)
Chest pain (General disorders) | 19 (22) | 9 (10)
Chills (General disorders) | 62 (267) | 13 (43)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (49) | 15 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (32) | 10 (14)
Erythema (Skin and subcutaneous tissue disorders) | 97 (625) | 24 (114)
Fatigue (General disorders) | 87 (504) | 32 (164)
Headache (Nervous system disorders) | 82 (369) | 24 (110)
Hospitalisation (Surgical and medical procedures) | 17 (24) | 7 (11)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 62 (271) | 20 (94)
Myalgia (Musculoskeletal and connective tissue disorders) | 90 (537) | 29 (132)
Nasopharyngitis (Infections and infestations) | 9 (12) | 4 (4)
Nausea (Gastrointestinal disorders) | 46 (174) | 18 (70)
Pain (General disorders) | 116 (947) | 36 (208)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 7 (7)
Pyrexia (General disorders) | 45 (120) | 8 (12)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Swelling (General disorders) | 91 (552) | 19 (69)
Vomiting (Gastrointestinal disorders) | 17 (33) | 10 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.